CLINICAL TRIAL: NCT02956434
Title: An Adjunctive Family Intervention for Individual PTSD Treatment
Brief Title: An Adjunctive Family Intervention for Individual Posttraumatic Stress Disorder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-013-16F; IK2CX001589 (NIH)
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Results first posted 2021-10-05 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Posttraumatic Neuroses
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief family intervention (Experimental): Participants will receive the BFI in this arm of the study. The BFI is a 2-session intervention for family members of Veterans who are beginning PTSD treatment.
  Interventions: Behavioral: Brief Family Intervention
- No intervention (No Intervention): Participants will not receive the BFI in this arm of the study. They will be eligible for any usual support or programming for the families of Veterans.

INTERVENTIONS:
Behavioral: Brief Family Intervention — Two 50-minute sessions aimed at helping family members be most supportive to their loved one's treatment goals.
  Arms: Brief family intervention

SUMMARY:
This study aims to test a brief family intervention (the BFI) to enhance individually-delivered PTSD treatment for Veterans.

DETAILED DESCRIPTION:
The investigators will enroll pairs of Veterans and one adult family member who lives with them. Veterans will be beginning a course of PTSD-focused treatment at the Boston VA; Veterans' treatment will not be limited or changed by their participation in this study.

Family members will receive or not receive (depending on which Phase of the study they are recruited in) the BFI. The BFI consists of 2 sessions in which the family member meets one-on-one with a clinician to discuss PTSD, PTSD treatment, and how families can be most helpful to patients in treatment.

Veterans and family members will also be interviewed about their opinions and experiences regarding family-inclusive treatment for PTSD. Clinicians will be recruited and enrolled to obtain their information and feedback (via qualitative interviews), and to deliver the intervention in Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Veterans must have a diagnosis of PTSD and be beginning a course of Prolonged Exposure (PE) or Cognitive Processing Therapy (CPT) at the Boston VA.
* Must also have an eligible family member who is willing to participate.

Exclusion Criteria:

* Current diagnosis of unstable bipolar disorder, substance dependence, past or present psychosis, or organic mental disorder
* Clear and current suicidal risk
* Current participation in family/couples therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Thompson-Hollands, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be released to other researchers as VA policy allows.
Supporting Information: Study Protocol, ICF
Time Frame: Entire study (baseline to 16 weeks)
Access Criteria: As per VA policy and local IRB approval

RESULTS

PARTICIPANT FLOW:
Groups:
- Brief Family Intervention - Veterans: The family members of these veterans will receive the BFI in this arm of the study. The BFI is a 2-session intervention for family members of Veterans who are beginning PTSD treatment.
  Brief Family Intervention: Two 50-minute sessions aimed at helping family members be most supportive to their loved one's treatment goals.
- No Intervention - Veterans: The family members of these veterans will not receive the BFI in this arm of the study. They will be eligible for any usual support or programming for the families of Veterans.
- Brief Family Intervention - Family Members: Participants will receive the BFI in this arm of the study. The BFI is a 2-session intervention for family members of Veterans who are beginning PTSD treatment.
  Brief Family Intervention: Two 50-minute sessions aimed at helping family members be most supportive to their loved one's treatment goals.
- No Intervention - Family Members: These family members will not receive the BFI in this arm of the study. They will be eligible for any usual support or programming for the families of Veterans.
Period: Overall Study
Arm/Group | Brief Family Intervention - Veterans | No Intervention - Veterans | Brief Family Intervention - Family Members | No Intervention - Family Members
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individuals (Veterans or family members) assigned to each group. The arms are paired -- the two Brief Family Intervention groups are paired dyad members, and the Usual-care CPT/PE Veterans and the No Intervention Family Members are also paired dyad members.
Groups:
- Brief Family Intervention - Veterans: Veterans will receive individually-delivered Cognitive Processing Therapy (CPT) or Prolonged Exposure (PE) to treat their PTSD.
  Their chosen family member will receive the BFI as an adjunctive treatment to the veteran's CPT/PE.
- Usual-care CPT/PE - Veterans: Veterans will receive individually-delivered Cognitive Processing Therapy (CPT) or Prolonged Exposure (PE) to treat their PTSD.
  Their chosen family member will NOT receive the BFI.
- Brief Family Intervention - Family Members: Family members will receive the BFI in this arm of the study. The BFI is a 2-session intervention for family members of Veterans who are beginning PTSD treatment.
  Brief Family Intervention: Two 50-minute sessions aimed at helping family members be most supportive to their loved one's treatment goals.
- No Intervention - Family Members: Participants will not receive the BFI in this arm of the study. They will be eligible for any usual support or programming for the families of Veterans.
- Total: Total of all reporting groups
Arm/Group | Brief Family Intervention - Veterans | Usual-care CPT/PE - Veterans | Brief Family Intervention - Family Members | No Intervention - Family Members | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.40 (18.12) | 38.70 (10.02) | 45.70 (17.25) | 38.30 (11.44) | 43.02 (14.852)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 10 | 10 | 20
  Male | 10 | 10 | 0 | 0 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 0 | 6
  White | 6 | 8 | 7 | 9 | 30
  More than one race | 2 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
CAPS-5 [Mean (Standard Deviation); unit: units on a scale] — Min value = 0, max value = 80. Higher scores mean worse outcome. Population: Only Veterans were administered the CAPS-5
  units on a scale
    number analyzed (Participants) | 10 | 10 | 0 | 0 | 20
    (all) | 37.80 (8.81) | 42.40 (8.81) |  |  | 40.10 (9.341)
SORTS [Mean (Standard Deviation); unit: units on a scale] — Min value = 0, max value = 112. Higher scores mean worse outcome. Population: Only family members completed the SORTS
  units on a scale
    number analyzed (Participants) | 0 | 0 | 10 | 10 | 20
    (all) |  |  | 33.30 (21.79) | 45.40 (27.24) | 39.35 (26.061)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale, 5th Edition
Description: A measure of PTSD severity and diagnostic status. Min value = 0, max value = 80. Higher scores mean worse outcome.
Time Frame: 16 weeks
Population: Only Veterans
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Family Intervention | No Intervention
Number analyzed (Participants) | 10 | 10
score on a scale | 18.60 (10.98) | 21.21 (9.91)

2. Primary Outcome: Treatment Attendance/Dropout
Description: A measure of Veterans' treatment attendance or premature dropout. Data represents the Veterans who dropped out of their standard-care PTSD treatment.
Time Frame: 16 weeks
Population: Only veterans
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Family Intervention | No Intervention
Number analyzed (Participants) | 10 | 10
Participants | 2 | 4

3. Secondary Outcome: Significant Others' Responses to Trauma Scale (SORTS)
Description: A measure of self-reported family accommodation of PTSD symptoms. Min value = 0, max value = 112. Higher scores mean worse outcome.
Time Frame: 16 weeks
Population: Only family members
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Family Intervention | No Intervention
Number analyzed (Participants) | 10 | 10
score on a scale | 22.82 (11.16) | 29.88 (24.87)

4. Secondary Outcome: Revised Dyadic Adjustment Scale
Description: A measure of relationship quality. Min value = 0, max value = 69. Higher scores mean better outcome.
Time Frame: 16 weeks
Population: Only family members
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Family Intervention | No Intervention
Number analyzed (Participants) | 10 | 10
score on a scale | 50.60 (8.38) | 51.00 (7.681)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: No difference in definitions
Arm/Group | Brief Family Intervention - Veterans | Usual-care CPT/PE - Veterans | Brief Family Intervention - Family Members | No Intervention - Family Members
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Family Intervention - Veterans (N=10) | Usual-care CPT/PE - Veterans (N=10) | Brief Family Intervention - Family Members (N=10) | No Intervention - Family Members (N=10)
Medication overdose (Psychiatric disorders) | 0 (0) | 1 (1) | NA | NA — Participant took more of their (non-study) psychiatric medication than was prescribed. No intervention was required.
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | NA | NA — Participant was involuntarily hospitalized following an aggressive episode

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT02956434/Prot_SAP_000.pdf